CLINICAL TRIAL: NCT02615106
Title: Phase 2 Study of Anti-angiogenetic Therapy With Radiotherapy for Pediatric Neuroblastoma
Brief Title: Anti-angiogenetic Therapy With Radiotherapy for Pediatric Neuroblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chuanying Zhu, doctor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SanghaiXinhua-001
Record Dates: First submitted 2015-11-22; First posted 2015-11-25 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Neuroblastoma
Keywords: Radiation Therapy; Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — endostar protein; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endostar Combined With Radiotherapy (Experimental): Drug: Endostar Endostar 7.5 mg/m2/day, day 1-14 Radiation: 21.6Gy/12Fx to the tumor bed and 36Gy/20Fx to the tumor
  Interventions: Drug: Endostar; Radiation: 21.6Gy/12Fx to the tumor bed and 36Gy/20Fx to the tumor

INTERVENTIONS:
Drug: Endostar — 7.5 mg/m2/day, day 1-14
  Other Names: recombinant human endostatin
Radiation: 21.6Gy/12Fx to the tumor bed and 36Gy/20Fx to the tumor — 21.6Gy/12Fx to the tumor bed and 36Gy/20Fx to the tumor

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Radiotherapy plus Endostar(Recombinant Human Endostatin) in patients with Pediatric Neuroblastoma.

DETAILED DESCRIPTION:
Clinical data proved that Endostar was a wild spectrum and safe antiangiogenesis factor which could suppress almost 65 kinds of tumor mass in animal models and affect about 12 percent human genome. So investigators design Radiotherapy plus Endostar to treat Pediatric Neuroblastoma to research the RR and safety. Investigators believe this treatment regimen may be a new approach to the pediatric neuroblastoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed neuroblastoma or ganglioneuroblastoma or elevated urinary catecholamine metabolites.
* Life expectancy of greater than 12 months.
* ECOG performance status ≤2
* Diagnostic Imaging MRI and/or CT of the area to be treated within 8 weeks of any treatment. Baseline bone marrow biopsy and bone scan (with 99mTc-diphosphonate or MIBG scan (131I-MIBG or 123I-MIBG) from time of original diagnosis is required.
* Because radiation is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability of the patient or the patient's legal guardian to understand and the willingness to sign a written informed consent document.
* Participants or their legal guardian must sign consent prior to the initiation of radiation therapy.

Exclusion Criteria:

* Patients will be ineligible if any prior therapeutic radiation therapy > 500 cGy has been delivered.
* Patients will be ineligible if chemotherapy was completed ≥ 1 year from the planned start date of radiation therapy or if the patient is referred for radiation therapy after a relapse following a regimen with chemotherapy alone.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Pregnant females are excluded. Women of childbearing age/menstruating must have a negative pregnancy test prior to initiation of radiation therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | first analysis will occur 1 month after accrual of all patients

SECONDARY OUTCOMES:
Progression free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Objective response rate (ORR) | first analysis will occur 1 month after accrual of all patients

CONTACTS AND LOCATIONS:
Overall Officials: mawei jiang, MD, Principal Investigator — The Department of Radiation Oncology, Xin Hua Hospital affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- The Department of Radiation Oncology, Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided